CLINICAL TRIAL: NCT03554941
Title: Non Invasive Vestibular Stimulation in Modulation of Vestibular and Balance Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, vghtpe user, Kao Chung-Lan, Taipei Veterans General Hospital, Taiwan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-12-004C
Record Dates: First submitted 2018-03-12; First posted 2018-06-13 (Actual); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Vestibular Insufficiency
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- noise stimulation (Experimental): noise stimulation
  Interventions: Device: noise stimulation

INTERVENTIONS:
Device: noise stimulation — noise stimulation

SUMMARY:
Background: Patients with bilateral vestibular hypofunction (BVH) frequently presented with dysequilibrium, dizziness and oscillopsia, leading to increased risk for fall. The mainstream for treatment of vestibular hypofunction remains to be vestibular rehabilitation, yet the effects can be limited in certain cases. Through the application of minimal amount of electrical stimulation, galvanic stimulation can induce polarization in the vestibular nerve, stimulating the saccule, utricle and semicircular canals within the vestibular apparatus. Galvanic stimulation has also been proven to activate cerebral cortex regions such as parieto-insular vestibular cortex (PIVC) and temporal-parietal junction area. It has been documented that vestibular stimulation with stochastic resonance could improve quiet stance stability in patients with vestibular hypofunction. The 3 dimensional effects of dynamic walking as well as the change of vestibular ocular reflex during stochastic resonance vestibular stimulation have never been discussed. Purposes: This 3-year project aims to investigate the effects of vestibular stimulation in VOR, static and dynamic stability, activation/connectivity of cerebral cortex and mechanisms of neuronal changes. Methods: First year the motion analysis and ICS head impulse video goggles were used to observe walking stability and eye movements in 30 healthy and 30 patients with BVH. In the second year, stochastic resonance vestibular stimulation will be applied to 30 healthy and 30 BVH individuals respectively. Using functional MRI, the changes of activated/deactivated areas in the cerebral cortex during stochastic resonance vestibular stimulation will be observed in both groups. In the third year, 60 BVH patients will be randomized into either sham or real vestibular stimulation group. Both groups will receive 3 times per week for 4 weeks of vestibular rehabilitation with exactly the same exercise protocols. SIRT1 related anti-aging genes will be analyzed through blood samples. Expected achievements: Combining safe stochastic resonance vestibular stimulation and exercises in this 3-year project, the neuroprotective mechanisms of vestibular exercises will be elucidated. The optimal strategy for vestibular rehabilitation can thus be established.

ELIGIBILITY:
Inclusion Criteria:

* vestibular insufficiency

Exclusion Criteria:

* 1. chronic diseases that may compromise vestibular function(eg. benign paroxysmal positional vertigo, post-traumatic vertigo, degenerative neural diseases, Whiplash injury), and patients with intracranial metal inplants or history of seizure
* 2. Patients with difficulty ambulation
* 3. Patients with cognitive function

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2017-07-20 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
deviation of center of gravity | Change from baseline afer 30 secs of stimulation
  deviation of center of gravity under each condition
motion analysis | Change from baseline afer 30 secs of stimulation
  step length
motion analysis | Change from baseline afer 30 secs of stimulation
  stride length
motion analysis | Immediately after 30 secs of stimulation
  trunk or pelvic rotation degree

SECONDARY OUTCOMES:
EEG(Electroencephalography) | Change from baseline after 30 secs of stimulation
  EEG to measured the change of brain activity
BOLD signal change assessed by functional MRI | Change from baseline afer 30 secs of stimulation
  Apply tDCS to stimulate brain and simultaneous fMRI exam，assess the neural activities change through BOLD signal

CONTACTS AND LOCATIONS:
Locations (1):
- TaipeiVGH, Taipei, Taiwan

REFERENCES:
- [Derived] Chen PY, Jheng YC, Wang CC, Huang SE, Yang TH, Hsu PC, Kuo CH, Lin YY, Lai WY, Kao CL. Effect of noisy galvanic vestibular stimulation on dynamic posture sway under visual deprivation in patients with bilateral vestibular hypofunction. Sci Rep. 2021 Feb 19;11(1):4229. doi: 10.1038/s41598-021-83206-z. PMID 33608568